CLINICAL TRIAL: NCT01105832
Title: Påskyndar PTH läkningen av Konservativt Behandlade Humerusfrakturer?
Brief Title: Does Teriparatide (rhPTH 1-34) Promote Fracture Healing in Proximal Humeral Fractures?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Torsten Johansson, MD, PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-017320-29
Record Dates: First submitted 2010-04-13; First posted 2010-04-19 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Humeral Fracture
Keywords: Teriparatide; fracture healing; proximal humeral fractures
MeSH Terms: conditions — Humeral Fractures; Shoulder Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proximal humeral fracture - intervention (Experimental): 20 patients will be randomized to 20 micrograms daily of Teriparatide (Forsteo)
  Interventions: Drug: Teriparatide
- Proximal humeral fracture (No Intervention): 20 patients will receive standard treatment (physiotherapy)

INTERVENTIONS:
Drug: Teriparatide — Teriparatide (Forsteo) 20 micrograms daily during four weeks
  Arms: Proximal humeral fracture - intervention

SUMMARY:
40 postmenopausal women, with a non-operated proximal humeral fracture, will be randomized to standard treatment (physiotherapy) or standard treatment + Forsteo (rhPTH 1-34) during 4 weeks. Follow-up will be at 7 weeks and 3 months including x-ray and DASH score (The Disabilities of the Arm, Shoulder and Hand) measuring physical function, and pain on a visual analoge scale (VAS).

Two doctors, blinded to the treatment, will judge the callus formation and healing on the x-rays and guess the treatment. The DASH score and the pain score will be compared between the treatment groups.

The investigators hypotheses are that callus formation and healing will be more pronounced and that patients have less pain and better function in the rhPTH 1-34 group.

ELIGIBILITY:
Inclusion Criteria:

* proximal humeral fracture
* postmenopausal woman 50 years or older
* non-surgical treatment

Exclusion Criteria:

* dementia or psychiatric disorder
* known malignancy < 5 years prior to fracture
* calcium above reference value
* signs of liver disease
* creatinine over ref. value
* inflammatory joint disease
* alcohol or drug abuse
* oral corticosteroid medication
* long-term NSAID-treatment (=> 3 months prior to fracture)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Callus formation and fracture healing at 7 weeks judged by a blinded assessor who will guess the treatment | 7 weeks

SECONDARY OUTCOMES:
Function | 7 weeks and 3 months
  The function in the upper extremity will be measured using DASH. The experimental group will be compared with the control group
Pain | 7 weeks and 3 months
  Pain at rest and during activity will be measured using a visual analogue scale (VAS). The experimental group will be compared with the control group

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Lasarettet i Motala, Motala
  - Department of Orthopaedics, Norrköping

REFERENCES:
- [Result] Aspenberg P, Genant HK, Johansson T, Nino AJ, See K, Krohn K, Garcia-Hernandez PA, Recknor CP, Einhorn TA, Dalsky GP, Mitlak BH, Fierlinger A, Lakshmanan MC. Teriparatide for acceleration of fracture repair in humans: a prospective, randomized, double-blind study of 102 postmenopausal women with distal radial fractures. J Bone Miner Res. 2010 Feb;25(2):404-14. doi: 10.1359/jbmr.090731. PMID 19594305
- [Result] Aspenberg P, Johansson T. Teriparatide improves early callus formation in distal radial fractures. Acta Orthop. 2010 Apr;81(2):234-6. doi: 10.3109/17453671003761946. PMID 20367417
- [Derived] Johansson T. PTH 1-34 (teriparatide) may not improve healing in proximal humerus fractures. A randomized, controlled study of 40 patients. Acta Orthop. 2016 Feb;87(1):79-82. doi: 10.3109/17453674.2015.1073050. Epub 2015 Jul 15. PMID 26179771